CLINICAL TRIAL: NCT04227808
Title: Safety and Efficacy of Lenvatinib as an Adjuvant Therapy in Patients With Hepatocellular Carcinoma Following Radical Resection: A Single-Arm and Open-Label Prospective Study
Brief Title: Efficacy and Safety of Lenvatinib as an Adjuvant Therapy for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Tongji Hospital (Other); Anhui Provincial Hospital (Other Government); West China Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Professor of Surgery, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-LEN-Adjuvant
Record Dates: First submitted 2020-01-05; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib Arm (Experimental): Experimental: Participants will be given lenvatinib (12 mg/d for body weight≥60kg, 8 mg/d for body weight < 60kg) for 12 months until disease recurrence or intolerance AEs or death.
  Interventions: Drug: Lenvima 4 mg Oral Capsule

INTERVENTIONS:
Drug: Lenvima 4 mg Oral Capsule — The participants will receive treatment with lenvatinib for 12 months after recruitment or until disease recurrence, intolerance AEs, or death. In case of treatment-related adverse effects, interruption or reduction is allowed.
  Other Names: Lenvatinib 4 mg Oral Capsule

SUMMARY:
Lenvatinib is the standard of care for patients with advanced hepatocellular carcinoma (HCC). The aim of the single-arm, open-label, phase II clinical trial is to evaluate the efficacy and safety of lenvatinib as an adjuvant therapy for patients underwent radical resection of HCC with a high risk of tumor recurrence.

Investigator hypothesize that lenvatinib may be an effective adjuvant treatment for HCC, and 12-month adjuvant treatment with lenvatinib can improve one-year recurrence-free survival rate (RFS) of HCC patients after surgical resection.

DETAILED DESCRIPTION:
There's no widely accepted adjuvant therapy for patients with HCC. Lenvatinib, a multi-targeted tyrosine kinase inhibitor, was approved for advanced or unresectable HCC. In this study, investigators aim to evaluate the effects and safety of adjuvant apatinib therapy for the patients who underwent curative resection for HCC with high risk of disease recurrence.

Participants who underwent radical resection for HCC with high risk of tumor recurrence will be recruited in this study. During 4 to 6 weeks after surgery, each participant will receive a screening visit to exclude residual tumors. Each eligible participant will be treated with lenvatinib until tumor recurrence, intolerant adverse effect, participant' refusal, or completing 12-month treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75;
2. Histological diagnosis of HCC;
3. Tumor stage before surgery: IIb/IIIa stage (>3 tumor nodules, or vascular invasion) HCC according to China Liver Cancer Staging System (or BCLC B/C/PVTT);
4. Underwent R0 resection (microscopic or macroscopic tumor clearance) in four to six weeks before recruitment; no residual tumor before recruitment by imaging study (MRI/CT), nor metastases to other organs;
5. Adequate liver, renal functions;
6. Written informed consent;
7. ECOG 0-1 and Child-Pugh A.

Exclusion Criteria:

1. WBC<4.0*10^9/L, HB<80 g/L, and PLT<75*10^9/L at blood screening;
2. Coagulation function: (prothrombin time) international normalized ratio (INR) >2.3, or extension of prothrombin time>6 seconds;
3. Liver function: serum albumin (ALB)<2.8 g/dl, total bilirubin (TBIL)>51.3μmol/L, alanine aminotransferase and aspartate aminotransferase (ALT and AST)>5 times the upper limit of normal range;
4. Renal function: serum creatinine (Cr)>1.5 times the upper limit of normal range;
5. lymph node metastases;
6. The participant has uncontrolled ascites, hepatic encephalopathy, Gilbert's syndrome, and sclerosing cholangitis, etc.;
7. The participant was included in other clinical trials 30 days before the selection;
8. Other conditions that the investigators considered that not unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
1-year RFS rate | 1 year after LPI
  1-year RFS rate is defined as the percentage of patients who do not experience tumor recurrence or death from any cause after 1-year treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  The duration from the date of first dosage to the date of death from any cause.
Adverse events | 13 months
  An adverse event (AE) refers to any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, but which does not necessarily have a causal relationship with this treatment. Number and classification of participants with treatment-related adverse events as assessed by CTCAE v4.0 were recorded.
Serious adverse events(SAE) | 13 months
  A serious adverse event (SAE) refers to an event in clinical trials that requires inpatient hospitalization or causes prolongation of existing hospitalization, permanent disability, incapacity, threats to life or death, and birth defect, etc. Number and classification of participants with treatment-related serious adverse events as assessed by CTCAE v4.0 were recorded.
Health-related quality of life | 13 months
  Health-related quality of life questionnaire measured by EORTC QLQ-HCC18.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (4):
- China (4):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Tongji Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - West China Hospital, Chengdu, Sichuan
  - 180 Fenglin Road, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Zhou J, Sun HC, Wang Z, Cong WM, Wang JH, Zeng MS, Yang JM, Bie P, Liu LX, Wen TF, Han GH, Wang MQ, Liu RB, Lu LG, Ren ZG, Chen MS, Zeng ZC, Liang P, Liang CH, Chen M, Yan FH, Wang WP, Ji Y, Cheng WW, Dai CL, Jia WD, Li YM, Li YX, Liang J, Liu TS, Lv GY, Mao YL, Ren WX, Shi HC, Wang WT, Wang XY, Xing BC, Xu JM, Yang JY, Yang YF, Ye SL, Yin ZY, Zhang BH, Zhang SJ, Zhou WP, Zhu JY, Liu R, Shi YH, Xiao YS, Dai Z, Teng GJ, Cai JQ, Wang WL, Dong JH, Li Q, Shen F, Qin SK, Fan J. Guidelines for Diagnosis and Treatment of Primary Liver Cancer in China (2017 Edition). Liver Cancer. 2018 Sep;7(3):235-260. doi: 10.1159/000488035. Epub 2018 Jun 14. PMID 30319983